CLINICAL TRIAL: NCT05756361
Title: A Family-Based Approach to Treat Obesity and Its Co-morbidities in Youth With Type 1 Diabetes (T1D) and Their Parents
Brief Title: Family-Based Treatment for Type 1 Diabetes
Acronym: FBT for T1D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Teresa Quattrin, Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006622: FBT for T1D; UL1TR001412 (NIH)
Record Dates: First submitted 2023-02-09; First posted 2023-03-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1; Obesity, Childhood; Overweight; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Pediatric Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 20 Child-Parent Dyads (Experimental): Family-Based Behavioral Treatment
  Interventions: Behavioral: Family-Based Treatment for T1D

INTERVENTIONS:
Behavioral: Family-Based Treatment for T1D — Our FBT curriculum, which has been delivered successfully in the specialty and primary care settings, has 3 components: 1. Meal planning including quality of carbohydrates and glycemic index for both parents and children while ensuring that youth have a balanced meal plan with adequate amounts of carbohydrates for optimal growth. Our FBT has a focus on "Food Literacy" including healthy food selection and sourcing of affordable healthy food, food preparation and preplanning, social engagement tailoring the meal plan to the needs to the family in socio cultural appropriate way and also feasibility based on logistics and economic aspects; 2. Physical activity (PA) component with shaping strategy to allow for a progressive shaping of easy PA starting, if needed, with as little as with 10 minutes of walking/day and strategies to incorporate PA in daily routines, family, and social activities; 3. Extensive behavioral component which has been shown to be very powerful in obesity treatment

SUMMARY:
Type 1 Diabetes carries high burden for affected youth and their families. Advances in insulin therapy and technology have been associated with increased obesity with 1/3 adolescents being overweight/obese. Since obesity runs in families and carries risk for poor outcomes psychologically and medically, the investigators are adapting our successful evidence-based Family Based Treatment for hybrid delivery to improve obesity and metabolic control in the affected youth and improve obesity and related co-morbidities in their parents.

DETAILED DESCRIPTION:
The investigators are conducting a 6-month (26 weeks) pilot trial enrolling 20 patients (6-17-year-old) with T1D and overweight/obesity and at least one parent with overweight/obesity and at least one associated co-morbidity, such as hypertension, pre-diabetes/T2D, or hyperlipidemia. The investigators realize that the age range chosen encompasses different developmental ages and are prepared to make some adaptations based on the intellectual and developmental abilities of the youth. For example, young children react very well to games related to food choices. Participants will have T1D duration >1 year (to exclude patients in the partial remission period), receive insulin therapy via pump or multiple daily injections, and wear a continuous glucose monitor. Both insulin regimens paired with continuous glucose monitor allow comparable potential to achieve optimal diabetes control. This study will test the feasibility of delivering an FBT intervention with a strong behavioral component to treat overweight in BOTH child and parent. The investigators will provide the participants with Body Trace Weight scales and instruct parents and youth to check their weight twice/week. The purpose of weight checking between in-person meetings is for the family coach to help the parent (and the child is old enough) relate weight changes to diet and activity habits/healthy behaviors and to develop plans to address weight gain relapse when needed. The choice of the Body Trace Weight scale is because it is a cellular enabled scale that will work even if there is a lapse in Wi-Fi availability and is user friendly without complicated set up procedures. Moreover, the investigators have already purchased them and will not need funding for them.

The intensity of the proposed schedule is in keeping with the treatment dose recommended by the United States Preventive Task Force recommendations. The coaching sessions will occur weekly for nine weeks (week 0,1,2,3,4,5,6, 7, 8), followed by sessions every two weeks for two months (wks. 10,12,14,16, 18), and then 2 sessions at a monthly interval (wks. 22 and 26). As described in the table below, the intensity of contact needs to be greater initially because this facilitates change in habits. However, "lack of time" is a major barrier to the acceptance of FBT programs for treatment of overweight and ultimately in the translation and dissemination of successful programs. Therefore, to overcome this barrier, after the initial four in person (IP) sessions, the investigators will alternate IP with virtual (V) meetings. Moreover, the investigators will coordinate the standard of care diabetes follow-ups (needed every 10-12 weeks) at the same time of the coaching sessions (IP + clinic at week 0-12 and 26).

Wk 0 1 2 3 4 5 6 7 8 10 12 14 16 18 22 26 IP+ CLINIC IP IP IP V IP V IP V V IP + CLINIC V IP V IP IP + CLINIC The coordination of the sessions with the standard of care visit will also involve the patient's diabetologist in following the patient's progress, providing positive feedback and learning from this program. From a practical standpoint, out of the 14 planned sessions, 6 will be virtual sessions, 3 will be in-person coordinated with the diabetes standard of care follow-up outpatient appointment, and seven would be in-person sessions. The investigators have experience with virtual delivery of FBT in the primary care setting during the COVID pandemic. Moreover, patients with T1D are accustomed to the use of digital health to upload their pump and sensors/glucose monitors. The investigators have conducted a 4-week pilot on the use of Wi-Fi scales in ten children 2-8 years old and their mothers (6/10 overweight or obese) who were instructed to monitor their weight and the child's weight twice week for a total of 8 times. 8/10 mothers monitored their weight and that of their child 7/8 times.

The investigators have considered the possibility of group sessions which foster learning and peer support and are cost-effective. Group education has been adopted especially in adults with T2D. While the investigators have conducted FBT group meetings in many instances in the past, they have been coupled with 1:1 meeting to tailor coaching to the particular needs of a participant and to "make up" missed group sessions. T1D is a chronic and very taxing disorder for patients and families. The coordination of group meetings imposes a "fixed day and time" regimen that cannot be met by many parents who need flexibility and tends to exclude single parents and those families who have health and socio-economic inequities, who could benefit the most from coaching. In the recently completed PLAN grant, a multicenter FBT implemented in the primary care setting the investigators adopted a 1:1 strategy which has allowed us to recruit 43% of minority families and 17% with income at the poverty line or below.

Our FBT curriculum, which has been delivered successfully in the specialty and primary care settings, has 3 components: 1. Meal planning including quality of carbohydrates and glycemic index for both parents and children while ensuring that youth have a balanced meal plan with adequate amounts of carbohydrates for optimal growth. Our FBT has a focus on "Food Literacy" including healthy food selection and sourcing of affordable healthy food, food preparation and preplanning, social engagement tailoring the meal plan to the needs to the family in socio cultural appropriate way and also feasibility based on logistics and economic aspects; 2. Physical activity (PA) component with shaping strategy to allow for a progressive shaping of easy PA starting, if needed, with as little as with 10 minutes of walking/day and strategies to incorporate PA in daily routines, family, and social activities; 3. Extensive behavioral component which has been shown to be very powerful in FBT for obesity and will be tailored to the needs of the patient with T1D. The program will focus on energy reduction, increased PA, and behavioral techniques to develop and sustain healthy habits conducive to reach healthy weight while balancing glycemic targets.

In the past, the investigators have compared the FBT intervention in a randomized fashion to an Education Control arm, where parents (and children if old enough) would receive education regarding meal planning and physical activity pertaining ONLY to the child (targeting child only) without a behavioral component and without treating the parent. This modality of controls for attention and still provides some benefit but not the same degree of weight loss. However, for this proposal, the investigators will deliver the treatment to 20 families without randomizing to a control arm because this is the first time the investigators are adapting our successful evidence based FBT for treatment of obesity in the general population to treat patients with T1D and obesity and their parents with obesity and related co-morbidities. Moreover, it is also the first time that the protocol (outside of pandemic constraints) includes a mix of in-person and virtual treatments. Therefore, with the limited time and funding, the investigators feel that the first step in this adaptation is to demonstrate that FBT to a new population using a hybrid program do work. The investigators propose, however, to compare the FBT intervention to a standard of care control group of patients matched for gender, age and HbA1c to the participants in this study. The investigators acknowledge that the major limitation of this control group is the fact that there is not randomization and also that the investigators will not be collecting parental data. Yet this, coupled with the change that each patient and parents will have compared to baseline, will give us some solid preliminary data to judge the effectiveness of the program and provide data for power calculations for extramural application supporting a randomized trial.

In contrast to Type 2 diabetes, T1D is not more prevalent in Black, Indigenous and People of Color (BIPOC). However, the highest rate of obesity in patients with T1D is indeed seen in patients with socio-economic disparities and minority status, and the investigators will prioritize enrollment of these patients. The investigators are aware of the inequities caused by the digital divide. The choice of cellular scales that enable communication during internet lapses was made to assist families who may have socio economic difficulties. The majority of these families still have cellular phones which will allow virtual contact. Therefore, the investigators will use some of the funds to help families with socio-economic disparities afford internet (if they do not have it) and a means to communicate electronically.

ELIGIBILITY:
Inclusion Criteria:

* T1D of 12 or more months duration
* Age 6-17-years
* Presence of overweight/obesity
* Youth uses a pump for insulin delivery and a continuous glucose monitoring device to monitor glycemic levels
* Youth has one parent with overweight/obesity willing to participate in the program

Exclusion Criteria:

* Child:

  * Chronic conditions other than T1D
  * Other autoimmune conditions other then T1D or autoimmune thyroiditis.
  * Medications that can affects weight, such as medications used to treat Attention Deficit Disorder or high dose steroids used to treat asthma.
  * Depression symptoms by standard of care Patient Health Questionnaire (PHQ) 9 in the child or parent
  * Inability to perform at least mild physical activity such as walking
  * Child with handicap (such as developmental delay or deafness) that would prevent him/her from benefitting from counseling in person and/or remotely Participating parent with
  * symptoms of depression assessed by standard of care PHQ
  * autoimmune disorders other than T1D or autoimmune thyroiditis
  * Participating parents with chronic disorder that is treated with medications that interfere with weight loss or are preventing him/her from performing at least mild physical activity

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Weight for parent and child | Baseline, 3 and 6 months
  Participants will be given Body Trace Weight Scales and will weigh themselves twice per week.

SECONDARY OUTCOMES:
Change in insulin dosing | baseline, 3 and 6 months
  Metrics will be obtained through Insulin pumps
In parents, change in severity of obesity co-morbidities | baseline, 3 and 6 months
  Participants will be given Body Trace Weight Scales and will weigh themselves twice per week. Parent co-morbidities will be tracked on a sheet
Change in HbA1c | baseline, 3 and 6 months
  Metrics will be obtained through Continuous Glucose Monitor
Change in time in range (TIR) - that is in optimal glycemic range | baseline, 3 and 6 months
  Metrics will be obtained through Continuous Glucose Monitor
In parents, change in medication dosing | baseline, 3 and 6 months
  Parent medications will be tracked on a sheet.

CONTACTS AND LOCATIONS:
Locations (1):
- Conventus, Buffalo, New York, United States